CLINICAL TRIAL: NCT04843163
Title: Examining the Impact of a Peer-Provided Psychoeducational Program for Parents: NAMI Basics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Sarah Kate Bearman, Study Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEAPLabUTNAMIBasics
Record Dates: First submitted 2021-04-05; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Mental Disorder, Child
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: Individuals are assigned to immediate NAMI Basics or waitlist control. Those in the waitlist control may take the NAMI Basics class after the 8 week waiting period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wave A (Immediate NAMI Basics) (Experimental): Once a participant has completed the questionnaires, that participant will be randomly assigned to either an immediate NAMI Basics class (Wave A), or an 8-week delay (Wave B) condition. Those in the immediate condition will be assigned to take the next available NAMI Basics class. Participants in both groups will be assessed at three time points. Participants in the immediate Basics group (Wave A) condition will be assessed pre-class, post-class, and 6 months after class has ended.
  Interventions: Behavioral: NAMI Basics
- Wave B (Waitlist Control) (No Intervention): Participants in the 8-week delay condition will be able to participate in a NAMI Basics class immediately following the 8-week time frame. Participants in the 8-week delay group (Wave B) will be assessed before the 8-week delay, after the 8-week delay (prior to their Basics course), and after the Basics course.

INTERVENTIONS:
Behavioral: NAMI Basics — NAMI Basics is a peer service program for caregivers of children with mental health needs. It was created by the National Alliance on Mental Illness (NAMI) and was adapted from their empirically supported model for caregivers of adult children with mental illness (Family-to-Family). The child-focused intervention, NAMI Basics, is a six-class curriculum focused on increasing caregiver knowledge about mental illness, empowering parents to advocate for their children across service systems, and introducing skills that assist in family problem-solving and communication (Brister et al., 2012). The program is currently available widely throughout the U.S. through certified trainers who volunteer with local NAMI affiliates and is provided free of charge to caregivers in a non-stigmatizing community setting (e.g., local school, church, community center). It is open to all caregivers, regardless of mental health diagnosis or time within a treatment system.
  Arms: Wave A (Immediate NAMI Basics)

SUMMARY:
This study will evaluate a peer service program for caregivers of youth struggling with mental illness using a program developed by the National Alliance on Mental Illness (NAMI) called NAMI Basics. This peer service program for caregivers was adapted from their successful and empirically supported model for caregivers of adult children with mental illness (Family-to-Family). The child-focused intervention, NAMI Basics, is a six-class curriculum focused on increasing caregiver knowledge about mental illness, empowering parents to advocate for their children across service systems, and introducing skills that assist in family problem-solving and communication.

The current study is a randomized effectiveness trial of NAMI Basics. Caregivers who are parenting youth with a mental illness (N = 175) referred to the NAMI Basics program through natural referral routes will be given the option to participate in the study, and if interested, randomly assigned to either an immediate NAMI Basics classes (Wave A) or an 8-week delay condition (Wave B), followed by initiation of the NAMI Basics class.

DETAILED DESCRIPTION:
This study will evaluate a peer service program for caregivers of youth struggling with mental illness using a program developed by the National Alliance on Mental Illness (NAMI) called NAMI Basics. This peer service program for caregivers was adapted from their successful and empirically supported model for caregivers of adult children with mental illness (Family-to-Family). The child-focused intervention, NAMI Basics, is a six-class curriculum focused on increasing caregiver knowledge about mental illness, empowering parents to advocate for their children across service systems, and introducing skills that assist in family problem-solving and communication. It is available widely throughout the U.S. through certified trainers who volunteer with local NAMI affiliates and is provided free of charge to caregivers in a non-stigmatizing community setting (e.g., local school, church, community center). It is open to all caregivers, regardless of mental health diagnosis or time within a treatment system. Families may be just beginning to recognize their child has a mental health challenge or may have been involved in service systems for many years. The program has been fully translated into Spanish, as well, and can be provided by Spanish-speaking trainers in many communities (known as Bases y Fundamentos de NAMI). NAMI Basics offers an inexpensive, non-stigmatizing strategy to increase families' access to information, training, and support in caring for their child with behavioral health challenges. The program can serve as an adjunct to traditional services or as a stand-alone program.

An initial pilot trial of NAMI Basics demonstrated pre-post increases in knowledge about youth mental illness and advocacy among a sample of 85 caregivers. A second study of 36 caregivers participating in NAMI Basics replicated and extended these results, demonstrating an increase in family empowerment and caregiver self-care, and reductions in inflammatory communication. However, more rigorous testing of the impact of the intervention, similar to that conducted with its "sister" program, needs to be conducted.

In order to more rigorously test the promising NAMI Basics program, we propose a randomized effectiveness trial. Caregivers who are parenting youth with a mental illness (N = 175) referred to the NAMI Basics program through natural referral routes will be given the option to participate in the study, and if interested, randomly assigned to either an immediate NAMI Basics classes (Wave A) or an 8-week delay condition (Wave B), followed by initiation of the NAMI Basics class. The NAMI Basics classes will be studied within five local NAMI affiliates in Texas. As the NAMI Basics program is translated and provided in Spanish, both Spanish and English classes will be run and evaluated as part of this research study.

ELIGIBILITY:
Inclusion Criteria:

* Any primary caregivers of youth (aged 2 to 18) with emotional or behavioral health problems referred to the NAMI Basics program via naturally occurring referral systems and who have signed informed consent for participation.
* Participants must be fluent in English or Spanish.

Exclusion Criteria:

* Only one caregiver per identified child (It may occur that two caregivers of the same child will enroll in the class and be interested in participating in the study. If two caregivers of the same child are enrolled in the class and interested in the research study, only one will complete study questionnaires. This will be determined by the caregivers themselves, and they will elect one reporter to complete study questionnaires.)
* Those who have attended 2 or more class sessions of NAMI Basics previously, at any point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Change in Parental Stress | Wave A: Baseline (Pre Intervention), 6 weeks - 8 weeks from class start (post intervention) ,and 6 month after class completion, Wave B: Baseline (Pre Intervention), 6 weeks (post waitlist), 12 weeks (directly after class completion)
  Parental Stress Scale (PSS). The PSS (Berry & Jones, 1995) is a self-report measure that assesses the level of stress experienced by caregivers and includes both positive and negative aspects of parenting. The measure is designed to assess changes in parental stress and changes in parenting capacity for parents who have access to services and targeted support. It consists of 18 items measured on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The items are statements about typical interactions with the child, both positive and negative, and caregivers must indicate the extent to which the agree or disagree with the statements.
Change in Parent Self-Competence, Expectancies, Efficacy, Knowledge, Self-Care | Wave A: Baseline (Pre Intervention), 6 weeks - 8 weeks from class start (post intervention) ,and 6 month after class completion, Wave B: Baseline (Pre Intervention), 6 weeks (post waitlist), 12 weeks (directly after class completion)
  Parent-Self-Competence Expectancies Efficacy Knowledge Self-Care (P-SEEKS). The PSEEKS (Olin, Kutash, & Hoagwood, N.d.) is a self-report measure that assesses parent self-efficacy and activation for parents of children with mental health needs. It is designed to capture changes in the area of self-efficacy for parents receiving targeted services or support. It includes measures across 6 domains: positive expectations about activation, self-competence, confidence and affirmation of parent role, self-care skills related to personal well-being, knowledge of formal mental health systems, knowledge of information networks and supports, and mental health services self-efficacy and the confidence to act. It consists of 31 items measured on 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree).
Change in Child Mental Health Symptoms | Wave A: Baseline (Pre Intervention), 6 weeks - 8 weeks from class start (post intervention) ,and 6 month after class completion, Wave B: Baseline (Pre Intervention), 6 weeks (post waitlist) , 12 weeks (directly after class completion)
  Youth Outcome Questionnaire (Burlingame, Wells, Hoag, et al., 2012; Y-OQ 2.01). The Y-OQ is a measure completed by caregivers to assess child treatment progress while receiving intervention. It is designed to be used with caregivers of children ages 4-17 and to capture total amount of distress experienced by the child. It consists of 64 items and caregivers must rate how frequently the described child behaviors occur. Rating options are: never or almost never, rarely, sometimes, sometimes, or always or almost always. The Y-OQ is published by OQ Measures and has been widely used in research studies.
Family Problem Solving and Communication | Wave A: Baseline (Pre Intervention), 6 weeks - 8 weeks from class start (post intervention) ,and 6 month after class completion, Wave B: Baseline (Pre Intervention), 6 weeks (post waitlist) , 12 weeks (directly after class completion)
  Family Problem Solving and Communication Scale. The Family Problem Solving and Communication Scale (McCubbin, McCubbin & Thompson, 1998) is a self-report measure used to assess family problem solving and communication style. It consists of 10 items, and caregivers must rate statements about their family's problem solving and communication style as False, Mostly False, Mostly True, or True.
Change in Mental Health Service Use | Wave A: Baseline (Pre Intervention), 6 weeks - 8 weeks from class start (post intervention) ,and 6 month after class completion, Wave B: Baseline (Pre Intervention), 6 weeks (post waitlist), 12 weeks (directly after class completion)
  The Short Service Assessment for Children and Adolescents- Brief (ShortSACA). The ShortSACA is a measure completed by an interviewer and caregivers to assess a child's use of mental health and social services. This includes the duration, type, frequency, and costs of services used, and includes both school-based and court-services. This tool has been widely used and studied (see Horowitz et al., 2001; Stiffman et al. 2000; Hoagwood et al., 2000). The ShortSACA is a shortened version of the full-length SACA and contains 30 items reflecting use of services over a period of time. This tool has been modified for this study to allow caregivers to complete the measure independently. The measure used for this study contains 28 items.
Change in Parent Attitudes Towards Psychological Services | Wave A: Baseline (Pre Intervention), 6 weeks - 8 weeks from class start (post intervention) ,and 6 month after class completion, Wave B: Baseline (Pre Intervention), 6 weeks (post waitlist) , 12 weeks (directly after class completion)
  Parent Attitudes Towards Psychological Services Inventory (PATPSI). The PATPSI (Turner, 2012) is a self-report measure that assesses caregiver attitudes towards outpatient mental health services. It measures help-seeking attitudes, intentions and mental health stigma. This measure consists of 26 items measured on a 5-point Likert scale ranging from 0 (strongly disagree) to 5 (strongly agree). (pre-intervention and post-intervention)

SECONDARY OUTCOMES:
Program Satisfaction | Wave A: 6-8 weeks after class start, Wave B: 12 weeks after randomization and immediately after NAMI Basics class
  NAMI Basics Program Evaluation. This measure assesses satisfaction with participation in the NAMI Basics course, solicits information from caregivers about how the program could be improved, and collects basic demographic information. It consists of 24 items total. The questionnaire includes 14 statements about the program and caregiver confidence in managing various situations. Caregivers are asked to rate these statements as on Likert-type scale from strongly agree to strongly disagree. The measure also includes 5 open-ended questions where caregivers are asked for their impression of the program, and any suggestion for improvement. Finally, the measure includes 5 questions which collect basic demographic information such as age, gender, race/ethnicity and how they were first referred to the NAMI Basics course.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kate Bearman, PhD, Principal Investigator — The University of Texas at Austin; Molly Lopez, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No